CLINICAL TRIAL: NCT02085616
Title: Smoking Cessation by Telephone. Effectiveness and Cost-effectiveness of Proactive and Reactive Services at the Swedish National Tobacco Quitline (SNTQ).
Brief Title: Effectiveness of the Swedish National Tobacco Quitline
Acronym: SNTQ
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis, revealed no additional effect of proactive over reactive service.
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other); Region Stockholm (Other Government); Västmanland County Council, Sweden (Other Government); Swedish Heart Lung Foundation (Other); Swedish Cancer Society (Other); The Swedish Research Council (Other Government); Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRL00-367
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Smoking Cessation; Tobacco Cessation
Keywords: Smoking cessation; Tobacco cessation; Quitline; Telephone counselling; Intensity
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation

ARMS (2):
- Proactive service (Experimental): Intervention: Tobacco cessation by telephone support. The structured treatment protocol is a mixture of motivational interviewing (MI), cognitive behaviour therapy, and pharmacological consultation. In the proactive service the callers to the quitline are offered a number of callbacks.
  Interventions: Behavioral: Proactive service
- Reactive service (Active Comparator): Intervention: Tobacco cessation by telephone support. The structured treatment protocol is a mixture of motivational interviewing (MI), cognitive behaviour therapy, and pharmacological consultation. In the reactive service the callers to the quitline are informed that they can themselves call back whenever they like.
  Interventions: Behavioral: Reactive service

INTERVENTIONS:
Behavioral: Proactive service — In the proactive service the callers to the quitline are offered a number of callbacks.
  Arms: Proactive service
Behavioral: Reactive service — In the reactive service the callers to the quitline are informed that they can themselves call back whenever they like.
  Arms: Reactive service

SUMMARY:
The purpose of this study was to compare the effectiveness of the high-intensity proactive service with the low-intensity reactive service at the Swedish National Tobacco Quitline (SNTQ). Our hypothesis was that the effectiveness is about 5% higher in proactive than in reactive service.

The structured treatment protocol is a mixture of motivational interviewing (MI), cognitive behavior therapy, and pharmacological consultation.The standard process at the SNTQ is to offer the client a choice of callback (proactive service) or no callback (reactive service). In the present study clients were not offered a choice, but were randomized to proactive service on even dates and to reactive service on odd dates. Data are collected through postal questionnaires, one baseline and one follow-up after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Tobacco users calling the SNTQ to discuss his/her own tobacco behaviour.
* The client gives verbal consent to sign up for cessation support.
* The client return a registration form including a baseline questionnaire

Exclusion Criteria:

* Snuff cessation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2009-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Point prevalence abstinence | 12 months
  Not a puff in the last week

SECONDARY OUTCOMES:
6-month continuous abstinence | 12 months
  Not a puff in the last 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gilljam, Prof, Principal Investigator — Karolinska Institutet; Ásgeir R Helgason, Assoc prof, Principal Investigator — Karolisnka Institutet; Eva Nohlert, PhD, Principal Investigator — Centre for Clinical Research Västerås, Uppsala University
Locations (3):
- Sweden (3):
  - Karolinska Institutet, Stockholm
  - Stockholm County Council, Stockholm
  - Centre for Clinical Research, Västerås

REFERENCES:
- [Derived] Nohlert E, Ohrvik J, Helgason AR. Self-perceived ability to cope with stress and depressive mood without smoking predicts successful smoking cessation 12 months later in a quitline setting: a secondary analysis of a randomized trial. BMC Public Health. 2018 Aug 28;18(1):1066. doi: 10.1186/s12889-018-5973-9. PMID 30153814
- [Derived] Nohlert E, Ohrvik J, Helgason AR. Effectiveness of proactive and reactive services at the Swedish National Tobacco Quitline in a randomized trial. Tob Induc Dis. 2014 Jun 3;12(1):9. doi: 10.1186/1617-9625-12-9. eCollection 2014. PMID 24936168